CLINICAL TRIAL: NCT04572217
Title: Medications After Adolescent Bariatric Surgery Protocol for Inadequate Weight Loss Following Sleeve Gastrectomy in Adolescents and Young Adults: A Pilot Feasibility Study
Brief Title: Medications After Adolescent Bariatric Surgery
Acronym: MAABS Protocol
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No available funding
Sponsor: Janey Pratt (Other)
Collaborators: Maternal and Child Health Research Institute (Unknown)
Responsible Party: Sponsor-Investigator, Janey Pratt, Clinical Associate Professor of Surgery, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54967; 1092951-100- KHAAX (Other Grant/Funding Number: MCHRI Clinical Fellowship Grant)
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Obesity
Keywords: Adolescent; Bariatric Surgery; Medications; Weight loss
MeSH Terms: conditions — Pediatric Obesity; Weight Loss | interventions — Topiramate; Phentermine

STUDY DESIGN:
Intervention Model Description: Pilot feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication Group (Experimental): Adolescent patients post vertical sleeve gastrectomy who have had inadequate weight loss, who consented for use of off-label medications prescribed at the discretion (one or both) of physician.
  Patients will be followed every 2-12 weeks over one year.
  All patients in this group will continue to follow the standard of care procedures of our multidisciplinary bariatric clinic, including frequent follow-up appointments, nutrition guidance, vitamin supplementation, exercise instruction, and healthy lifestyle education.
  Interventions: Drug: Topiramate; Drug: Phentermine
- Non-Medication Group (No Intervention): Adolescent patients post vertical sleeve gastrectomy who had inadequate weight loss and did not consent for use of off-label medications.
  All patients in this group will continue to follow the standard of care procedures of our multidisciplinary bariatric clinic, including frequent follow-up appointments, nutrition guidance, vitamin supplementation, exercise instruction, and healthy lifestyle education.

INTERVENTIONS:
Drug: Topiramate — Topiramate (starting dose 25 mg daily, max dose 100 mg daily)
  Arms: Medication Group
Drug: Phentermine — Phentermine (starting dose 8 mg, max dose 16 mg)
  Arms: Medication Group

SUMMARY:
This study will assess the feasibility to assess practicality of early weight loss medication usage in adolescent patients post-VSG with inadequate weight loss. Participants who enroll in the study will be prescribed off-label use of weight loss medications for a period of up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients in the LPCH/Stanford bariatric and weight management clinics
* Inadequate weight loss after vertical sleeve gastrectomy

Exclusion Criteria:

* Adequate weight loss after surgery;
* Unwilling to consent or adhere to safety monitoring plan;
* Any life-threatening or terminal diseases
* Currently pregnant, breastfeeding, or thinking of becoming pregnant
* Allergy or medical contraindication to phentermine or topiramate;
* History of drug or alcohol abuse;
* No known medication interactions;
* Significant renal or hepatic impairment;
* Participation in a study of an investigational medication 30 days prior to screening, while the patient is on study, and for 30 days after their last dose of study treatment

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who are able to consent for off-label medication use as a measure of feasibility | Up to 1 year

SECONDARY OUTCOMES:
Average daily rate of compliance with medication administration | Up to 1 year
Percent change from baseline in % BMI | Baseline (initiation of medication), 1 year
Type of weight loss medication prescribed | Up to 1 year
  Type of weight loss medication prescribed, according to type and dose
Number of participants experiencing side effects | Up to 1 year
Timing of the implementation of off-label medications after vertical sleeve gastrectomy | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Janey Pratt, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldenkamp AP, Baker G, Mulder OG, Chadwick D, Cooper P, Doelman J, Duncan R, Gassmann-Mayer C, de Haan GJ, Hughson C, Hulsman J, Overweg J, Pledger G, Rentmeester TW, Riaz H, Wroe S. A multicenter, randomized clinical study to evaluate the effect on cognitive function of topiramate compared with valproate as add-on therapy to carbamazepine in patients with partial-onset seizures. Epilepsia. 2000 Sep;41(9):1167-78. doi: 10.1111/j.1528-1157.2000.tb00322.x. PMID 10999556
- [Background] Boyer EW, Shannon M. The serotonin syndrome. N Engl J Med. 2005 Mar 17;352(11):1112-20. doi: 10.1056/NEJMra041867. No abstract available. PMID 15784664
- [Background] Chanoine JP, Richard M. Early weight loss and outcome at one year in obese adolescents treated with orlistat or placebo. Int J Pediatr Obes. 2011 Apr;6(2):95-101. doi: 10.3109/17477166.2010.519387. Epub 2010 Sep 22. PMID 20858149
- [Background] Czepiel KS, Perez NP, Campoverde Reyes KJ, Sabharwal S, Stanford FC. Pharmacotherapy for the Treatment of Overweight and Obesity in Children, Adolescents, and Young Adults in a Large Health System in the US. Front Endocrinol (Lausanne). 2020 May 13;11:290. doi: 10.3389/fendo.2020.00290. eCollection 2020. PMID 32477270
- [Background] Doose DR, Wang SS, Padmanabhan M, Schwabe S, Jacobs D, Bialer M. Effect of topiramate or carbamazepine on the pharmacokinetics of an oral contraceptive containing norethindrone and ethinyl estradiol in healthy obese and nonobese female subjects. Epilepsia. 2003 Apr;44(4):540-9. doi: 10.1046/j.1528-1157.2003.55602.x. PMID 12681003
- [Background] Hendricks EJ, Srisurapanont M, Schmidt SL, Haggard M, Souter S, Mitchell CL, De Marco DG, Hendricks MJ, Istratiy Y, Greenway FL. Addiction potential of phentermine prescribed during long-term treatment of obesity. Int J Obes (Lond). 2014 Feb;38(2):292-8. doi: 10.1038/ijo.2013.74. Epub 2013 May 17. PMID 23736363
- [Background] Kramer CK, Leitao CB, Pinto LC, Canani LH, Azevedo MJ, Gross JL. Efficacy and safety of topiramate on weight loss: a meta-analysis of randomized controlled trials. Obes Rev. 2011 May;12(5):e338-47. doi: 10.1111/j.1467-789X.2010.00846.x. Epub 2011 Mar 28. PMID 21438989
- [Background] Lewis KH, Fischer H, Ard J, Barton L, Bessesen DH, Daley MF, Desai J, Fitzpatrick SL, Horberg M, Koebnick C, Oshiro C, Yamamoto A, Young DR, Arterburn DE. Safety and Effectiveness of Longer-Term Phentermine Use: Clinical Outcomes from an Electronic Health Record Cohort. Obesity (Silver Spring). 2019 Apr;27(4):591-602. doi: 10.1002/oby.22430. PMID 30900410
- [Background] Ahamada Safna Mariyam M, Sen S, Vijayan K. Topiramate: Safety in migraine patients. J Young Pharm. 2013 Mar;5(1):30-1. doi: 10.1016/j.jyp.2012.12.001. Epub 2013 Mar 6. No abstract available. PMID 24023450
- [Background] Martin R, Kuzniecky R, Ho S, Hetherington H, Pan J, Sinclair K, Gilliam F, Faught E. Cognitive effects of topiramate, gabapentin, and lamotrigine in healthy young adults. Neurology. 1999 Jan 15;52(2):321-7. doi: 10.1212/wnl.52.2.321. PMID 9932951
- [Background] Rich S, Rubin L, Walker AM, Schneeweiss S, Abenhaim L. Anorexigens and pulmonary hypertension in the United States: results from the surveillance of North American pulmonary hypertension. Chest. 2000 Mar;117(3):870-4. doi: 10.1378/chest.117.3.870. PMID 10713017
- [Background] Rissanen A, Lean M, Rossner S, Segal KR, Sjostrom L. Predictive value of early weight loss in obesity management with orlistat: an evidence-based assessment of prescribing guidelines. Int J Obes Relat Metab Disord. 2003 Jan;27(1):103-9. doi: 10.1038/sj.ijo.0802165. PMID 12532161